CLINICAL TRIAL: NCT01244945
Title: Effect of Lactobacillus Reuteri DSM 17938 on Gut Motility in Patients With Functional Constipation
Brief Title: Lactobacillus Reuteri DSM 17938 in Functional Constipation
Acronym: LRFC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Francesco Russo, MD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1026D
Record Dates: First submitted 2010-11-17; First posted 2010-11-22 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Functional Constipation
Keywords: Functional Constipation; Functional Foods; Probiotics; Lactobacillus reuteri

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L. reuteri DSM 17938 (Experimental)
  Interventions: Dietary Supplement: L. reuteri DSM 17938
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Group

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938 — L. reuteri will be administered at 1x10^8 CFU dosage in form of tabs. In order to ensure colonization (run in), 4 tabs will be administered per os daily (4x10^8CFU/die) for 15 days. Then administration will continue with 2 tabs daily (2x10^8 CFU/die) for 90 days.
  Arms: L. reuteri DSM 17938
Other: Placebo Group — Placebo tabs identical in form, taste and consistency to active tabs
  Arms: Placebo

SUMMARY:
The diffusion of gastrointestinal (GI) chronic diseases is significantly increased during the last century in western countries. In the USA and Northern Europe, constipation is twofold the prevalence found in the East and Southern Europe. In Italy, constipation affects up to 15-17% of the whole adult population. Of them, more than half (about 10%) treats this disorder by assuming laxatives, while the remaining does not even assume drugs. A close relationship between intestinal environment and bacterial flora has been found. As a matter of fact changes in the intestinal physiology can modify the composition of bacterial flora as well as modifications in the intestinal microbiota can modify the physiology of the gut. The probiotic effects on the GI motility can be due to substances released by bacteria and/or products of their fermentation. Also, probiotic may indirectly act by the release of neuroendocrine factors and/or substances released by the immune system. Clinically, it has already been demonstrated that probiotics exert a positive effect on symptoms and intestinal habit in constipated IBS patients. In this framework, the idea to perform a long lasting intervention study in patients with functional constipation treated with probiotics sounds convincing. The present study is a randomized, double blind, placebo controlled, monocentric study, concerning the evaluation of efficacy of 3 months administration of Lactobacillus reuteri DSM 17938 in patients with functional constipation, as defined by the Rome criteria. Clinical, physiological, hematological and immunologic variables will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilment of the Rome Criteria III for functional constipation
* Availability of at least one GI imaging study during the last five years (colonoscopy, sigmoidoscopy, abdominal ultrasound, barium enema)
* Commitment to availability for the whole study period

Exclusion Criteria:

* Major abdominal surgery
* Presence of any concomitant diseases such as organic GI diseases and/or lactose and gluten intolerance; medical or psychiatric illness
* Alarming symptoms (rectal bleeding, weight loss, etc)
* Family history of peptic ulcer, colorectal cancer, or IBD
* Abnormal laboratory data or thyroid function.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Improvement in gastrointestinal symptoms after 3 months of probiotic administration | Before the start of the study (Time 0) and after 90 days of treatment (Time 90)
  Validated and structured questionnaires to evaluate gastrointestinal symptoms, to confirm functional constipation diagnosis and to exclude IBS variant constipation. Score of gastrointestinal symptoms with Gastrointestinal Symptom Rating Score (GSRS); Constipation Symptom Score (CSS); Constipation QoL, Constipation Rome criteria, Diary for the symptoms and for intestinal behavior. These questionnaires will be administered at baseline, after 45 days of treatment, and at the end of treatment.

SECONDARY OUTCOMES:
Changes in metabolic parameters after 3 months of probiotic administration | Before the start of the study (time 0) and after 90 days of treatment (Time 90)
  Lipidic and glucidic profile; evaluation of circulating immunological parameters, short chain fatty acid (SCFA)faecal concentrations. The evaluations will be performed at baseline, after 45 days of treatment and at the end of treatment.
Changes in physiological parameters after 3 months of probiotic administration | Before the start of the study (Time 0) and after 90 days of treatment (Time 90)
  Physiological parameters: Quali/Quantitative evaluation of the colonic transit time (TTC) with radiopaque markers (qualitative study : RX after 3 days from the 20 markers assumption. Quantitative study: RX after 3 days from the assumption of 10 markers a day for 6 days in patients with TTC delayed), non invasive evaluation of gastric electrical activity and gastric emptying time (cutaneous electrography (EGG) and 13C octanoic acid breath test). The evaluations will be performed at baseline, after 45 days of treatment and at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Riezzo, M.D., Principal Investigator — Azienda Ospedaliera Specializzata in Gastroenterologia IRCCS "Saverio de Bellis"
Locations (1):
- National Institute for Digestive Diseases IRCCS "S. de Bellis", Castellana Grotte, Bari, Italy

REFERENCES:
- [Background] Indrio F, Riezzo G, Raimondi F, Bisceglia M, Cavallo L, Francavilla R. The effects of probiotics on feeding tolerance, bowel habits, and gastrointestinal motility in preterm newborns. J Pediatr. 2008 Jun;152(6):801-6. doi: 10.1016/j.jpeds.2007.11.005. Epub 2007 Dec 26. PMID 18492520
- [Background] Russo F, Clemente C, Linsalata M, Chiloiro M, Orlando A, Marconi E, Chimienti G, Riezzo G. Effects of a diet with inulin-enriched pasta on gut peptides and gastric emptying rates in healthy young volunteers. Eur J Nutr. 2011 Jun;50(4):271-7. doi: 10.1007/s00394-010-0135-6. Epub 2010 Oct 12. PMID 20938778
- [Background] Riezzo G, Clemente C, Leo S, Russo F. The role of electrogastrography and gastrointestinal hormones in chemotherapy-related dyspeptic symptoms. J Gastroenterol. 2005 Dec;40(12):1107-15. doi: 10.1007/s00535-005-1708-7. PMID 16378174
- [Background] Riezzo G, Chiloiro M, Russo F. Functional foods: salient features and clinical applications. Curr Drug Targets Immune Endocr Metabol Disord. 2005 Sep;5(3):331-7. doi: 10.2174/1568008054863790. PMID 16178793
- [Background] Valerio F, Russo F, de Candia S, Riezzo G, Orlando A, Lonigro SL, Lavermicocca P. Effects of probiotic Lactobacillus paracasei-enriched artichokes on constipated patients: a pilot study. J Clin Gastroenterol. 2010 Sep;44 Suppl 1:S49-53. doi: 10.1097/MCG.0b013e3181d2dca4. PMID 20495470